CLINICAL TRIAL: NCT02466711
Title: A Single-center, Placebo-controlled, Double-blind Study to Evaluate the Effect of Relamorelin on Satiation, Gastric Volume, Gastric Accommodation and Distal Gastric Function in Healthy Volunteers
Brief Title: Effect of Relamorelin on Satiation, Gastric Volume, Gastric Accommodation and Distal Gastric Function in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Motus Therapeutics, Inc. (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RM-131-010
Record Dates: First submitted 2015-06-05; First posted 2015-06-09 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Gastric Motility
Keywords: gastric motility
MeSH Terms: interventions — relamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relamorelin (Active Comparator)
  Interventions: Drug: Relamorelin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Relamorelin — Double blind RM-131 will be delivered three times by injection during the course of the study
  Other Names: RM-131
  Arms: Relamorelin
Drug: Placebo — Double blind Placebo will be delivered three times by injection during the course of the study
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of relamorelin (RM-131) on gastric volume, motor and sensory effects in healthy patients.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent prior to any study procedures, and be willing and able to comply with study procedures
2. No medical problems or chronic diseases, specifically, no type 2 diabetes mellitus
3. Body mass index of 18-35 kg/m²
4. Female subjects must have negative urine pregnancy tests and must not be lactating prior to receiving study medication and radiation exposure. For females able to bear children, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study. Female subjects unable to bear children must have this documented in the medical record (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]).

Exclusion Criteria:

1. Unable or unwilling to provide informed consent or to comply with study procedures
2. Diagnosis of gastrointestinal diseases
3. Structural or metabolic diseases that affect the GI system
4. Unable to avoid the following over- the- counter medications 48 hours prior to the baseline period and throughout the study:

   1. Medications that alter GI transit including laxatives, magnesium and aluminum containing antacids, prokinetics, erythromycin,
   2. Analgesic drugs including NSAIDs and COX-2 inhibitors NOTE: stable doses of thyroid replacement, estrogen replacement, low-dose aspirin for cardioprotection, and birth control (but with adequate backup contraception as drug-interactions with birth control have not been conducted) are permissible.
5. History of recent surgery (within 60 days of screening)
6. Acute or chronic illness or history of illness, which in the opinion of the Investigator, could pose a threat or harm to the subject or obscure interpretation of laboratory test results or interpretation of study data such as frequent angina, Class III or IV congestive heart failure, moderate impairment of renal or hepatic function, poorly controlled diabetes, etc.
7. Any clinically significant abnormalities on physical examination or laboratory abnormalities identified in the medical record, as determined by the Investigator
8. Acute GI illness within 48 hours of initiation of the baseline period
9. Females who are pregnant or breastfeeding
10. History of excessive alcohol use or substance abuse
11. Participation in an investigational study within the 30 days prior to dosing in the present study
12. Any other reason, which in the opinion of the Investigator, would confound proper interpretation of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Gastric volume measured by single photon emission computed tomography (SPECT) | Measured during the 1 hour study procedure
  Calculation of gastric volume by single photon emission computed tomography (SPECT)
Satiety measured by the Hunger/Satiety questionnaire | Measured during a 1 hour study procedure
  Measurement of satiety by completion of the Hunger/Satiety questionnaire after ingesting a nutrient drink
Gastric motility measured by gastroduodenal manometry | Measured during the 4 hour study procedure
  Measurement of gastric motility by gastroduodenal manometry

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic - Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Nelson AD, Camilleri M, Acosta A, Busciglio I, Linker Nord S, Boldingh A, Rhoten D, Ryks M, Burton D. Effects of ghrelin receptor agonist, relamorelin, on gastric motor functions and satiation in healthy volunteers. Neurogastroenterol Motil. 2016 Nov;28(11):1705-1713. doi: 10.1111/nmo.12870. Epub 2016 Jun 9. PMID 27283792